CLINICAL TRIAL: NCT05970406
Title: Effects of High Intensity Dysphagia Rehabilitation on Adults With Dysphagia s/p Acute Ischemic Stroke in an Acute Rehab Facility
Brief Title: High Intensity Dysphagia Rehab for Acute Ischemic Stroke Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00335053
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Dysphagia Following Cerebrovascular Accident

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Participants in high intensity dysphagia therapy (Experimental): Participants with acute dysphagia who will receive high intensity dysphagia therapy during stay in inpatient rehab facility
  Interventions: Other: high intensity dysphagia therapy

INTERVENTIONS:
Other: high intensity dysphagia therapy — Intensive swallowing interventions with Speech Language Pathologists to begin within 24 hours of video swallow study results. Daily treatment will include two 30-minute sessions, 5-6 days a week which will include the evidence-based dysphagia exercises focusing on tongue resistance, head lift/chin tuck against resistance and expiratory muscle strength training tasks

SUMMARY:
The purpose of this study is to determine a standardized protocol for swallowing therapy and this protocol's effects on recovery after a stroke

DETAILED DESCRIPTION:
This study will include adults, aged 18-99, who are admitted to Johns Hopkins Bayview (JHBMC) Rehabilitation Unit following an acute ischemic stroke with a diagnosis of dysphagia, determined by instrumental assessment with a Video Fluoroscopic Swallowing Study (VFSS). All participants will be asked to complete an informed consent form prior to admission to the study. Initial objective assessment of swallowing with video fluoroscopic swallowing assessment will be completed within 72 hours of admission to the unit. Participants with PAS scores of greater than or equal to 3 and FOIS scores of less than or equal to 6 will be admitted to the study and asked to complete the Eating Assessment Tool (EAT-10) score sheets. Intensive swallowing interventions with Speech Language Pathologists will begin within 24 hours. Daily treatment will include two 30-minute sessions, 5-6 days a week which will include the evidence-based dysphagia exercises focusing on tongue resistance, head lift/chin tuck against resistance and expiratory muscle strength training tasks. Devices utilized will include the Iowa Oral Performance Instrument (IOPI), and the Positive Expiratory Pressure (PEP) Respironics device or the Expiratory Muscle Strength Training (EMST150) device. Each session will involve IOPI measurements of lingual strength with endurance tasks set at 60% and 75% max strength scores to be completed for total of 10 attempts at each level for isometric and isokinetic tasks; Expiratory muscle strength training with EMST150 or PEP Respironics (dependent on strength levels) will be set at 75% max resistance levels per training method, for 25 completions per session; Shaker or Chin Tuck Against Resistance (CTAR) using 4.5 inch standard rubber ball - determined by patient positioning restrictions or tolerance- will be completed with goals of isometric hold for 1 minute x3 attempts and isokinetic x10 x3 attempts each session. At least one session per day will include consumption of ice chips and/or food dependent on PAS levels. At least one additional VFSS will be completed prior to discharge from study, as is standard of care within the JHBMC Rehab Unit. Outcome measures will be assessed with pre and post PAS scores (comparing initial and final VFSS results), EAT 10 scores and FOIS scores as well as documented improvements in IOPI and EMST/PEP levels at two-week intervals and will continue throughout the acute comprehensive inpatient rehabilitation unit (ACIR) stay as indicated. A follow up phone call with each participant will occur between 4-6 weeks post discharge from the and be completed with EAT-10 and FOIS over phone by Speech Language Pathologists or the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18-99
2. Ischemic Stroke
3. Identified to have acute dysphagia s/p ischemic stroke
4. Able to follow 1-step commands for swallowing directions

Exclusion Criteria:

1. Younger than 18, older than 100
2. Hemorrhagic Stroke, Subarachnoid hemorrhage, subdural hematoma, epidural hematoma
3. h/o dysphagia
4. Advanced progressive neurological disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with improved swallowing as assessed by the improved Penetration Aspiration Scale (PAS) | up to 6 weeks
  Measured with improved Penetration Aspiration Scale (PAS)
Number of participants with improved swallowing as assessed by the Functional Oral Intake Scale (FOIS) | up to 6 weeks
  Measured with the Functional Oral Intake Scale (FOIS)
Number of participants with perceived improvements in swallowing | up to 6 weeks
  Measured with improved EAT-10 Questionnaire Scores

CONTACTS AND LOCATIONS:
Overall Officials: Alba M Azola, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Buchholz DW. Dysphagia associated with neurological disorders. Acta Otorhinolaryngol Belg. 1994;48(2):143-55. PMID 8209677
- [Background] Buchholz DW. Oropharyngeal dysphagia due to iatrogenic neurological dysfunction. Dysphagia. 1995 Fall;10(4):248-54. doi: 10.1007/BF00431417. PMID 7493505
- [Background] Lugger KE. Dysphagia in the elderly stroke patient. J Neurosci Nurs. 1994 Apr;26(2):78-84. doi: 10.1097/01376517-199404000-00005. PMID 8077779
- [Background] Mann G, Hankey GJ, Cameron D. Swallowing disorders following acute stroke: prevalence and diagnostic accuracy. Cerebrovasc Dis. 2000 Sep-Oct;10(5):380-6. doi: 10.1159/000016094. PMID 10971024
- [Background] Martino R, Foley N, Bhogal S, Diamant N, Speechley M, Teasell R. Dysphagia after stroke: incidence, diagnosis, and pulmonary complications. Stroke. 2005 Dec;36(12):2756-63. doi: 10.1161/01.STR.0000190056.76543.eb. Epub 2005 Nov 3. PMID 16269630
- [Background] Gonzalez-Fernandez M, Ottenstein L, Atanelov L, Christian AB. Dysphagia after Stroke: an Overview. Curr Phys Med Rehabil Rep. 2013 Sep;1(3):187-196. doi: 10.1007/s40141-013-0017-y. PMID 24977109
- [Background] Krekeler BN, Rowe LM, Connor NP. Dose in Exercise-Based Dysphagia Therapies: A Scoping Review. Dysphagia. 2021 Feb;36(1):1-32. doi: 10.1007/s00455-020-10104-3. Epub 2020 Mar 5. PMID 32140905
- [Background] Malandraki GA, Rajappa A, Kantarcigil C, Wagner E, Ivey C, Youse K. The Intensive Dysphagia Rehabilitation Approach Applied to Patients With Neurogenic Dysphagia: A Case Series Design Study. Arch Phys Med Rehabil. 2016 Apr;97(4):567-574. doi: 10.1016/j.apmr.2015.11.019. Epub 2015 Dec 19. PMID 26711168
- [Background] Burkhead LM, Sapienza CM, Rosenbek JC. Strength-training exercise in dysphagia rehabilitation: principles, procedures, and directions for future research. Dysphagia. 2007 Jul;22(3):251-65. doi: 10.1007/s00455-006-9074-z. Epub 2007 Apr 25. PMID 17457549
- [Background] Alkhuwaiter M, Davidson K, Hopkins-Rossabi T, Martin-Harris B. Scoring the Penetration-Aspiration Scale (PAS) in Two Conditions: A Reliability Study. Dysphagia. 2022 Apr;37(2):407-416. doi: 10.1007/s00455-021-10292-6. Epub 2021 Apr 21. PMID 33880656
- [Background] Crary MA, Mann GD, Groher ME. Initial psychometric assessment of a functional oral intake scale for dysphagia in stroke patients. Arch Phys Med Rehabil. 2005 Aug;86(8):1516-20. doi: 10.1016/j.apmr.2004.11.049. PMID 16084801
- [Background] Belafsky PC, Mouadeb DA, Rees CJ, Pryor JC, Postma GN, Allen J, Leonard RJ. Validity and reliability of the Eating Assessment Tool (EAT-10). Ann Otol Rhinol Laryngol. 2008 Dec;117(12):919-24. doi: 10.1177/000348940811701210. PMID 19140539
- [Background] Balou M, Herzberg EG, Kamelhar D, Molfenter SM. An intensive swallowing exercise protocol for improving swallowing physiology in older adults with radiographically confirmed dysphagia. Clin Interv Aging. 2019 Feb 11;14:283-288. doi: 10.2147/CIA.S194723. eCollection 2019. PMID 30804667